CLINICAL TRIAL: NCT06124248
Title: RISE Intervention: Heading to Sustainable Movement Behavioural Change in People with Stroke
Brief Title: Effectiveness of the RISE Intervention
Acronym: RISE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, Martijn F. Pisters, PhD, PT, Principal Investigator, UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL83940.000.23; RAAK.PRO04.093 (Other Grant/Funding Number: SIA RAAK PRO); 10930012310010 (Other Grant/Funding Number: ZonMw)
Record Dates: First submitted 2023-10-13; First posted 2023-11-09 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Sedentary Behaviour; Stroke
Keywords: Physical activity; Cardiovascular diseases; Sedentary time; Sitting time; Movement behaviours; Behaviour change; Sedentary behaviour; Stroke; Secondary prevention; Costs; Cost analysis; Cost effectiveness; MACE; Prevention
MeSH Terms: conditions — Stroke; Motor Activity; Cardiovascular Diseases; Sedentary Behavior

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The investigator who carries out the T1 follow-up measurement (end of the intervention period), will be blinded for treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): RISE intervention and usual care
  Interventions: Behavioral: RISE intervention
- Control group (No Intervention): Usual care

INTERVENTIONS:
Behavioral: RISE intervention — The RISE intervention: a 15-weeks blended behavioral intervention, where a primary care physiotherapist coaches participants on striking the balance in their 24h activity pattern, with a focus on reducing and interrupting their sedentary time. This will subsequently lead to an increase in physical activity. Next to that, insights into their personal sleep pattern, sleep hygiene rules and advices will be provided.
  Primary care physiotherapists coach people with a first-ever stroke in their home setting by using behavior change techniques and the RISE eCoaching system. The RISE eCoaching system consists of 1) an activity monitor, 2) a smartphone application that provides real-time feedback and contains e-learning modules, 3) a monitoring dashboard for the physiotherapist. Participants receive participatory support from someone from their social network (e.g., partner or close friend) who joins them in the intervention.
  Arms: Experimental group

SUMMARY:
Study aim:

Primarily, to investigate the effectiveness of the RISE blended behaviour change intervention in people with a first stroke to prevent major adverse cardiovascular events (i.e., recurrent stroke or TIA, acute coronary events and cardiovascular death, MACE) after 1 year follow-up compared to standard care, and cost-effectiveness. For this aim, 376 persons are enrolled in the experimental group and 376 in the control group. Considering loss to follow up, it is expected that around 950-1000 patients need to be included during baseline measurement in total.

Additionally, to determine the effectiveness of the RISE intervention on reducing sedentary behaviour after discharge from acute hospital care in community dwelling people with a first-ever stroke, who have a sedentary movement behavioural pattern (so called 'sedentary prolongers' and 'sedentary movers') in comparison to usual care, at the end of the intervention period (T1). For this aim, 59 persons are enrolled in the experimental group and 59 in the control group. Considering loss to follow up, it is expected that around 197 patients need to be included during baseline measurement in total.

Who can participate? People aged over 18, who return home after acute care with a first-ever stroke, who are independent in walking with or without a walking aid, will be included in the RISE intervention study.

What does the study involve? In this clinical randomized controlled trial, participants with first-ever stroke and a sedentary movement pattern will be included and randomly assigned to either the experimental group who will receive RISE intervention and usual care or the control group who will receive usual care. Primary and secondary outcome will be measured at baseline, post-treatment and six, nine and 12 months post-randomisation.

DETAILED DESCRIPTION:
Rationale: People who have suffered a stroke are at high risk of functional decline, recurrent stroke and premature mortality. High amounts of sedentary behaviour, accumulated in prolonged bouts and low amounts of moderate to vigorous physical activity increase the risk of cardiovascular disease. Based on earlier research it is expected that a healthier balance in the 24h activity pattern (sedentary time, physical activity and sleep) reduces the risk of a second cardiovascular event. To support patients with stroke to strike the balance in their 24h activity pattern, a behavioural change coaching intervention focusing on reducing and interrupting their sedentary time was designed. A pilot study has been performed, and the RISE intervention seems feasible in reducing sedentary behaviour in people after stroke.

Objective: To determine the effectiveness of the RISE intervention on preventing major adverse cardiovascular effects (MACE), after discharge from acute hospital care in community dwelling people after first-ever stroke, who have a sedentary movement behavioural pattern. In addition, the effects on 24h activity pattern, cost-effectiveness, and usability of the RISE intervention will be investigated.

Study design: In this clinical randomized controlled trial, participants with first-ever stroke and a sedentary movement pattern will be included and randomly assigned to either the experimental group who will receive RISE intervention and usual care or the control group who will receive usual care. Primary and secondary outcomes will be measured at baseline, post-treatment (four months), and six, nine, and 12 months post-randomisation.

Study population: People aged over 18, who return home after acute care with a first-ever stroke, who are independent in walking with or without a walking aid, will be included in the RISE intervention study.

Intervention (if applicable): Participants will receive the RISE intervention, a 15-weeks blended behavioural intervention, where a primary care physiotherapist coaches participants on striking the balance in their 24h activity pattern, with a focus on reducing and interrupting their sedentary time. This will subsequently lead to an increase in physical activity. Next to that, insights into their personal sleep pattern, sleep hygiene rules and advices will be provided. Primary care physiotherapists coach people with a first-ever stroke in their home setting by using behaviour change techniques and the RISE eCoaching system. The RISE eCoaching system consists of 1) an activity monitor, 2) a smartphone application that provides real-time feedback and contains e-learning modules, 3) a monitoring dashboard for the physiotherapist. Participants receive participatory support from someone from their social network (e.g., partner or close friend) who joins them in the intervention (see image 1).

Participants in the control group receive usual care, according to hospital specific guidelines.

Main study parameters/endpoints: Effectiveness of RISE intervention on preventing major adverse cardiovascular events.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The burden and risk of participating in the RISE intervention are considered low. The participants will receive a blended coaching intervention to reduce and interrupt their sedentary behaviour. The blended intervention includes ten face-to-face or online sessions of a primary care physiotherapist, wearing an activity monitor during the intervention period, and support from the smartphone application. During the intervention people will be encouraged to sit less and move more. The participant will participate in a baseline and post intervention measurements. This includes wearing an activity monitor, questionnaires and performing physical tests. All measurements are non-invasive. Participants can shower and perform all other daily activities while wearing the activity monitor. The other measurements will take about 3.5 hours in total, and will be carried out online or at people&amp;amp;amp;amp;#39;s homes. Included participants are physically capable of performing these physical activities and are coached by a physiotherapist. Therefore, the risk involved in participating is low. Additional burden of the intervention is low since visits of the physiotherapist will be at home or online

The possible benefits of participating in the study are: 1) insights in own movement behaviour and 2) (if someone is randomized to the RISE intervention group) the RISE intervention may help to reduce sedentary time, which may lower the risk on recurrent stroke.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in the baseline measurement of the intervention study, a subject must meet all of the following criteria:

1. Aged 18 years or older;
2. All types of first-ever stroke diagnosed in hospital within six months before start of the RISE intervention;
3. Able to walk independently, as defined by a Functional ambulation categories score of at least 3;
4. Independent regarding activities of daily living pre-stroke, as defined by a Barthel Index score of >18;
5. Discharged to the home-setting;
6. Not participating in a physical rehabilitation program lasting ≥ 3 months;
7. Given their written informed consent.

Exclusion Criteria:

A potential subject will be excluded from participation in this study if:

1. The participant has insufficient knowledge or is cognitively unable to understand the Dutch language of the intervention content;
2. The participant has severe comorbidities that withhold that person from safely reducing and interrupting their sedentary time (e.g. sever pulmonary diseases, hart failure or malignity's) as determined with the Physical Activity Readiness Questionnaire;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2023-11-29 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Cardiovascular Events (MACE) | T1 (3 months), T2 (6 months), T3 (9 months), T4 (12 months)
  MACE, a composite of clinical end points of recurrent stroke or Transcient Ischaemic Attack (TIA) (definition in American Heart Association guidelines (44)), acute coronary events, and cardiovascular death. Stroke recurrence will be diagnosed by acute neurological symptoms and signs, and confirmed by magnetic resonance imaging. Acute coronary events (myocardial infarction (MI), cardiac revascularization, hospitalization with unstable angina) are diagnosed according to Consensus Conference of the European College of Cardiology and American College of Cardiology criteria (45). Deaths are regarded to be attributable to a cardiovascular cause (fatal MI, fatal stroke (i.e. death within 1 month of MI or stroke), sudden death caused by definite coronary artery disease, congestive heart failure) unless a non-cardiac death could be confirmed. This information about MACE will be collected at T1, T2, T3 and T4 using patient records from general practitioners and a questionnaire to participants.

SECONDARY OUTCOMES:
Cost-Effectiveness | T0 (baseline), T1 (3 months), T2 (6 months), T3 (9 months), T4 (12 months)
  Assessed for MACE and quality adjusted life years (QALYs). QALYs will be based on the patients' responses to EQ 5D-5L (46). These responses will be converted into utility values using the Dutch tariff , after which QALYs will be estimated using linear interpolation between measurement points (47). All costs related to the RISE intervention will be considered: costs of intervention, other healthcare, informal care, sports, unpaid productivity, absenteeism, and presenteeism costs. Intervention costs will be micro-costed, meaning that detailed data will be gathered about the number and kinds of resources are used while providing the RISE intervention as well as information about their respective unit costs. All other costs will be measured at T0-T4 using modified versions of the iMTA Medical Consumption Questionnaire (iMCQ) and the iMTA Productivity Cost Questionnaire (iPCQ) (48). In accordance with the Dutch manual for costing studies in health care
Quality of life | T0 (baseline), T1 (3 months), T2 (6 months), T3 (9 months), T4 (12 months)
  Health Related Quality of Life will be measured with the EuroQol-5D (EQ-5D) (50, 51) at T0, T1, T2, T3 and T4. This questionnaire comprises of 5 dimensions i.e., mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Per dimension, patients are asked to indicate their health status on a 5-point Likert scale (1 = no problems; 5 = extreme problems). The health states can be converted into utility units by means of the Dutch rates (52). Utilities represent quality of life into a single number that ranges from 0 (death) to 1 (full health). Quality Adjusted Life Years (QALY's) can subsequently be calculated by multiplying the patients' utilities by the duration of time they spent in that particular health status.
Patients' healthcare utilization and patients' (unpaid) productivity losses | T1 (3 months), T2 (6 months), T3 (9 months), T4 (12 months)
  Patients' healthcare utilization and patients' (unpaid) productivity losses will be measured using cost questionnaires.
  There will be made use of retrospective 3-month cost questionnaires (at T1, T2, T3 and T4) to avoid recall bias. Healthcare utilization will be valued using Dutch standards costs (56). If these are unavailable, prices reported by professional organizations will be used. will be valued in accordance with the "Dutch Manual of Costing".
24-hour movement behaviour (sedentary behaviour, physical activity, sleep) | T0 (baseline), T1 (3 months), T2 (6 months), T4 (12 months)
  24-hour movement behaviour consists of movement behaviour (sedentary time and physical activity) and sleep. 24-hour movement behaviour is measured with the ActivPAL (PAL Technologies Ltd, Glasgow, United Kingdom) at T0, T1, T2 and T4 (34). This monitor is combination of a triaxial accelerometer and inclinometer, worn on the anterior side of the unaffected thigh, and detects if someone is either sedentary (sitting, lying or reclining), standing or walking. The ActivPAL is sealed in a waterproof sleeve and attached to the skin using hypoallergic tape. Participants are instructed to wear the ActivPAL for eight consecutive days. The first 24 hour of the data will be removed in order to counteract a possible Hawhorne effect (53). This ActivPAL is reliable (Intraclass correlation coefficient 0.79-0.99) and valid (98-100% accuracy) for measuring sedentary time and posture transitions during daily life in people with stroke (41-43).

OTHER OUTCOMES:
Safety during the RISE intervention and follow-up measurements. | T0 (baseline), T1 (3 months), T2 (6 months), T3 (9 months), T4 (12 months)
  Safety will be objectified by the number of adverse events registered by the researcher during the intervention and/or during the follow-up measurements following the registration process (T0, T1, T2, T3, T4).
Physical functioning and participation | T0 (baseline), T1 (3 months)
  Physical functioning and participation, measured with the Short Physical Performance Battery (SPPB) at T0 and T1. THE SPPB is an objective assessment tool for evaluating lower extremity functioning in older persons, which gives insight in someone's walking speed, balance and leg strength. The SPPB consists of a balance test, a gait speed test and a chair stand test, of which each item is score with 1, 2 or 4 points. The maximal total score is 12, in which a higher score indicates better lower extremity functioning. The SPPB has an excellent interrater reliability (Intraclass Correlatin Coefficient (ICC) = 0.81 to 0.91) and excellent test-retest reliability (ICC = 0.84). (54, 55). The validity of the SPPB for measuring lower extremity function is moderate to high (0.66-0.79) (56).
Sleep quality and quantity | T0 (baseline), T1 (3 months), T2 (6 months), T4 (12 months)
  Sleep quality and quantity, measured with Emfit sleep tracker, at T0, T1, T2 and T4. The Emfit QS sleep tracker (Emfit Ltd, Vaajakoski, Finland; 542 3 70 3 1.4 mm) has recently been validated in healthy adult participants using an electrocardiography based reference device. The Emfit QS showed good validity and reliability in measuring heart rate during the sleep period (57). Next to the Emfit QS, experienced sleep quality is measured with the Pittsburgh Sleep Quality Index (PSQI). The PSQI is a 19-item self-reported questionnaire about experienced sleep quality in the past month. The PSQI shows a structural validity ranging between 0.70 and 0.83 (58).
Fatigue | T0 (baseline), T1 (3 months), T2 (6 months), T4 (12 months)
  Level of fatigue, is according to the Stroke Recovery Roundtable on fatigue, measured with the Fatigue Severity Scale-7 (FSS-7) and Visual Analogue Scale at T0, T1, T2 and T4. The items are asked about the past few weeks and relate to the perceived severity offatigue in different daily situations. The FSS-7 measures chronic fatigue in 7 items with a 7-point likert scale (ranging from 'totally disagree' to 'totally agree'). The final score is the mean of the 7 item scores. A final score of ≥4 indicates that the severity of fatigue has a medium to high impact on daily life. The FSS-7 demonstrates excellent item-reliability (Cronbach's alpha 0.87-0.93) in measuring change in fatigue over time (59).
Stroke physical impact | T0 (baseline), T1 (3 months), T2 (6 months), T4 (12 months)
  Stroke physical impact will be assessed using the Stroke Impact Scale (SIS) physical at T0, T1, T2 and T4. This questionnaire has 37 questions in 5 domains (strength, hand function, activities daily living /Instrumental activities daily living, mobility and participation/ role and function). In this study, the domain 'activities daily living' is used. These questions are answered on a 5-point Likert scale ranging from 1, negative (e.g. 'no strength at all' or 'extremely difficult'), to 5 (e.g. 'a lot of strength' or 'not difficult at all'). The SIS shows excellent internal consistency with Cronbach alpha ranging from 0.80 to 0.95. The test-retest reliability was investigated with reported Intraclass Correlation Coefficients (ICC) ranging from 0.70 to 0.94 (60).
Walking speed | T0 (baseline), T1 (3 months)
  Walking speed will be determined using the 5 meter walk test (5MWT) at T0 and T1, in which the participants is asked to walk 5 meters 3 times. Form the average duration of these three times the walking speed is calculated in meters per second (63, 64). The 5MWT has a standardized responsive mean of 1.2 (64)
Self-efficacy | T0 (baseline), T1 (3 months), T2 (6 months), T4 (12 months)
  Self-efficacy, measured with the self-efficacy for symptom management scale (SESx) at T0, T1, T2 and T4. The Self-Efficacy for Symptom Management Scale (SESx) will be used to assess self-efficacy. This questionnaire consists of 13 items scored on a 10-point scale ranging from 'not confident at all' to 'completely confident'. A higher score indicating higher self-efficacy (68).
Self-management skills | T0 (baseline), T1 (3 months), T2 (6 months), T4 (12 months)
  Self-management skills, measured with Patient Activation Measure (PAM) at T0, T1, T2 and T4. Patient self-management skills are assessed by the Dutch version of the short form Patient Activation Measure (PAM 13-Dutch) (69, 70). The PAM 13-Dutch is a reliable 13-item instrument and assesses patient (or consumer) self reported knowledge, skills and confidence for self-management of one's health or chronic condition. The answering categories per item are 4-point Likert scales, ranging from totally disagree to totally agree and 'non applicable'. A higher score (range 1-100) indicates a higher level of self-management.
Compliance to the RISE intervention | T1 (3 months)
  Compliance to the treatment protocol will be measured with a questionnaire filled out by the physical therapists at T1. Compliance consists of 1) the number of people that completed the intervention (with and without missing sessions); 2) The number of participants that mist one or more of the face to face sessions, the reasons for missing, and the percentage of missed sessions per participant; 3) The amount of sessions the participatory support was present; 4) The average amount of times participants used the RISE eCoaching system per week
End-user satisfaction, feasibility and acceptability | T1 (3 months)
  With the End-User Computing Satisfaction (EUCS) and Post-Study System Usability Questionnaire (PSSUQ) and System Usability Scale (SUS) at T1. The EUCS is a 12-item questionnaire to measure end-use computing satisfaction of the (experimental group) participant and physiotherapists about usage of the RISE eCoaching system. All items are scored with a 5-point Likert scale ('almost never' to 'almost always').The PSSUQ is a 19-item instrument that assesses the perceived satisfaction of a user with a system, in this case the RISE eCoaching system. The PSSUQ has an overall reliability score of 0.97. The SUS is a questionnaire that measures the perceived usability of the m-health part of the intervention by posing 10 statements which the participant can rate on a 5-points Likert scale ('completely agree' to 'completely disagree'). The score ranges from 0-100, with a higher score indicating a higher perceived usability. It is a reliable (0.85) instrument to measure participants perceived usa
Mental health status | T0 (baseline), T1 (3 months), T2 (6 months), T4 (12 months)
  Mental health status will be measured with the Hospital Anxiety and Depression Scale (HADS) at T0, T1, T2 and T4.
  The HADS is a short questionnaire of 14 items with a 4-point Likert scale. A higher score indicates more mental health problems.
Patient characteristics | T0 (baseline), T1 (3 months)
  Patient characteristics will be obtained (age, gender, education level, living situation (number of persons in the household), comorbidities, measured with CIRS (50), stroke characteristics (type of stroke, side of stroke, time since stroke) and vascular risk factors (coronary artery disease, AF, diabetes, hypertension, clinical obesity, smoking and alcohol use, hyperlipidemia) with an intake questionnaire (case report form) at T0. Cognitive functioning will be assessed using the Montreal Cognitive Assessment (MoCA). MoCA assesses eight domains of cognitive functioning with small tasks. The scores range from 0-30, a score of less than 26 indicates impaired cognitive function (53).Vascular risk factors will be measured with a questionnaire at T0, accompanied by measuring Body Mass Index (BMI) and blood pressure as risk factors for a cardiovascular event at T0, T1.

CONTACTS AND LOCATIONS:
Overall Officials: Martijn F Pisters, Dr., Principal Investigator — UMC Utrecht Brain Center and Fontys University of Applied Sciences
Locations (21):
- Netherlands (21):
  - Fysio 4 Den Bosch, 's-Hertogenbosch, North Brabant
  - Meras & Vital Fysiotherapie, Eersel, North Brabant
  - PMC Eindhoven, Eindhoven, North Brabant
  - Stroomz Prinsejagt, Eindhoven, North Brabant
  - Fysiotherapie Zesgehuchten, Geldrop, North Brabant
  - JVDI De Fysioclub, Helmond, North Brabant
  - Fysiotherapie Rakthof, Helmond, North Brabant
  - Vivent, Rosmalen, North Brabant
  - Van Hoof, centrum voor therapie en gezondheid, Valkenswaard, North Brabant
  - Fysio Annette de Gooijer, Vlijmen, North Brabant
  - Fysiofit Vught, Vught, North Brabant
  - Fysio Vught Noord, Vught, North Brabant
  - Fysiotherapie Beelen, Breukelen, Utrecht
  - Fysiotherapie Zorgspectrum Houten eerstelijn, Houten, Utrecht
  - Fysiotherapie Groene Biezen, IJsselstein, Utrecht
  - MTCFysio, Mijdrecht, Utrecht
  - Leidsche Rijn Julius Gezondheidscentra, Utrecht, Utrecht
  - Rembrandt fysiotherapie en revalidatie, Veenendaal, Utrecht
  - Fysio Frankenhof, Wijk bij Duurstede, Utrecht
  - Synergy Fysiotherapie, Woerden, Utrecht
  - Van Tongeren Fysiotherapeuten, Zeist, Utrecht

IPD SHARING:
Plan to Share IPD: Yes
Pseudonymized data will be available upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: As soon as all data have been collected and analyzed, individual participant data (IPD) will be shared upon reasonable request.
Access Criteria: No access restrictions.

REFERENCES:
- [Derived] Biemans CFM, Hartman YAW, Broers S, Pagen S, Hendrickx W; RISE Study Group; van Dongen JM, Verschuren OW, English C, Veenhof C, Visser-Meily JMA, Pisters MF. Secondary prevention by striking the balance in 24-hour movement behaviour by empowering people at risk with a stroke: rationale and design of the RISE intervention randomised controlled trial. BMJ Open. 2025 Jun 5;15(6):e094894. doi: 10.1136/bmjopen-2024-094894. PMID 40473286